CLINICAL TRIAL: NCT00090584
Title: Behavior Enhances Drug Reduction of Incontinence
Brief Title: Behavior Enhances Drug Reduction of Incontinence (BE-DRI)
Acronym: BE-DRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE-DRI (completed)
Record Dates: First submitted 2004-08-27; First posted 2004-08-31 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-05

CONDITIONS: Urinary Incontinence (UI)
Keywords: Urge urinary incontinence (UUI); Drug/Behavior treatment
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge | interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination therapy (Experimental): Women randomly assigned to this condition receive 10 weeks of anti-cholinergic medication (tolterodine) and behavioral training.
  Interventions: Drug: Tolterodine; Behavioral: Behavioral training
- Drug therapy alone (Active Comparator): Women assigned to this arm received 10 weeks of anti-cholinergic medication (tolterodine), only.
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Tolterodine — 4mg/d for 10 weeks. Could be reduced to 2mg/d for managing side effects.
Behavioral: Behavioral training — Training in pelvic floor muscle control and exercises; behavioral strategies to diminish urgency, suppress bladder contractions and prevent incontinence; delayed voiding; and individualized fluid management.
  Arms: Combination therapy

SUMMARY:
The primary aim of this study is to test if the addition of behavioral treatment to drug therapy for the treatment of urge incontinence will increase the number of patients who can discontinue drug therapy and sustain a significant reduction of incontinence.

ELIGIBILITY:
Inclusion:

* Female
* Urge predominant incontinence
* Incontinent > 3 mos
* Available for 8 mos of followup

Exclusion:

* Pregnancy or < 6 mos post-partum
* Hypersensitivity to drug (tolterodine)
* Systemic disease that affects bladder function (e.g., Parkinson's disease, Multiple Sclerosis, spinal cord injury)
* History of extensive behavior treatment

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2004-08; Primary Completion 2005-12 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Steers, M.D., Study Chair — University of Virginia
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Oakwood Hospital and Medical Center, Royal Oak, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Urinary Incontinence Treatment Network (UITN). Design of the Behavior Enhances Drug Reduction of Incontinence (BE-DRI) study. Contemp Clin Trials. 2007 Jan;28(1):48-58. doi: 10.1016/j.cct.2006.06.002. Epub 2006 Jun 18. PMID 16919506
- [Background] Borello-France D, Burgio KL, Goode PS, Markland AD, Kenton K, Balasubramanyam A, Stoddard AM; Urinary Incontinence Treatment Network. Adherence to behavioral interventions for urge incontinence when combined with drug therapy: adherence rates, barriers, and predictors. Phys Ther. 2010 Oct;90(10):1493-505. doi: 10.2522/ptj.20080387. Epub 2010 Jul 29. PMID 20671098
- [Background] Brubaker L, Lukacz ES, Burgio K, Zimmern P, Norton P, Leng W, Johnson H, Kraus S, Stoddard A. Mixed incontinence: comparing definitions in non-surgical patients. Neurourol Urodyn. 2011 Jan;30(1):47-51. doi: 10.1002/nau.20922. PMID 21181960
- [Background] Burgio KL, Kraus SR, Borello-France D, Chai TC, Kenton K, Goode PS, Xu Y, Kusek JW; Urinary Incontinence Treatment Network. The effects of drug and behavior therapy on urgency and voiding frequency. Int Urogynecol J. 2010 Jun;21(6):711-9. doi: 10.1007/s00192-010-1100-x. Epub 2010 Feb 9. PMID 20143047
- [Background] Burgio KL, Kraus SR, Menefee S, Borello-France D, Corton M, Johnson HW, Mallett V, Norton P, FitzGerald MP, Dandreo KJ, Richter HE, Rozanski T, Albo M, Zyczynski HM, Lemack GE, Chai TC, Khandwala S, Baker J, Brubaker L, Stoddard AM, Goode PS, Nielsen-Omeis B, Nager CW, Kenton K, Tennstedt SL, Kusek JW, Chang TD, Nyberg LM, Steers W; Urinary Incontinence Treatment Network. Behavioral therapy to enable women with urge incontinence to discontinue drug treatment: a randomized trial. Ann Intern Med. 2008 Aug 5;149(3):161-9. doi: 10.7326/0003-4819-149-3-200808050-00005. PMID 18678843
- [Background] Fitzgerald MP, Lemack G, Wheeler T, Litman HJ; Urinary Incontinence Treatment Network. Nocturia, nocturnal incontinence prevalence, and response to anticholinergic and behavioral therapy. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Nov;19(11):1545-50. doi: 10.1007/s00192-008-0687-7. Epub 2008 Aug 14. PMID 18704249
- [Background] Goode PS, Burgio KL, Kraus SR, Kenton K, Litman HJ, Richter HE; Urinary Incontinence Treatment Network. Correlates and predictors of patient satisfaction with drug therapy and combined drug therapy and behavioral training for urgency urinary incontinence in women. Int Urogynecol J. 2011 Mar;22(3):327-34. doi: 10.1007/s00192-010-1287-x. Epub 2010 Oct 13. PMID 20945064
- [Background] Markland AD, Richter HE, Kenton KS, Wai C, Nager CW, Kraus SR, Xu Y, Tennstedt SL; Urinary Incontinence Treatment Network. Associated factors and the impact of fecal incontinence in women with urge urinary incontinence: from the Urinary Incontinence Treatment Network's Behavior Enhances Drug Reduction of Incontinence study. Am J Obstet Gynecol. 2009 Apr;200(4):424.e1-8. doi: 10.1016/j.ajog.2008.11.023. Epub 2009 Feb 6. PMID 19200939
- [Background] Richter HE, Burgio KL, Chai TC, Kraus SR, Xu Y, Nyberg L, Brubaker L. Predictors of outcomes in the treatment of urge urinary incontinence in women. Int Urogynecol J Pelvic Floor Dysfunct. 2009 May;20(5):489-97. doi: 10.1007/s00192-009-0805-1. Epub 2009 Jan 30. PMID 19183825
- [Background] Zimmern P, Litman HJ, Mueller E, Norton P, Goode P; Urinary Incontinence Treatment Network. Effect of fluid management on fluid intake and urge incontinence in a trial for overactive bladder in women. BJU Int. 2010 Jun;105(12):1680-5. doi: 10.1111/j.1464-410X.2009.09055.x. Epub 2009 Nov 13. PMID 19912207
- [Background] Fitzgerald MP, Dubeau CE, Kraus SR, Johnson HW Jr, Rahn DD, Mallett V, Stoddard AM, Zyczynski HM; Urinary Incontinence Treatment Network. Patient expectations did not predict outcome of drug and behavioral treatment of urgency urinary incontinence. Female Pelvic Med Reconstr Surg. 2011 Sep;17(5):231-7. doi: 10.1097/SPV.0b013e31822dd10b. PMID 22453106
- [Background] Dyer KY, Xu Y, Brubaker L, Nygaard I, Markland A, Rahn D, Chai TC, Stoddard A, Lukacz E; Urinary Incontinence Treatment Network (UITN). Minimum important difference for validated instruments in women with urge incontinence. Neurourol Urodyn. 2011 Sep;30(7):1319-24. doi: 10.1002/nau.21028. Epub 2011 May 11. PMID 21563210
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598
- See also: www.uitn.net — http://www.uitn.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July, 2004 and January, 2006 4,043 women were screened for eligibility and 561 provided written consent. After further screening, 134 were found to be ineligible, 119 withdrew consent and 1 was excluded erroneously. The remaining 307 were randomized to one of the treatment arms.
Pre-assignment Details: Of the 134 found to be ineligible after consent, for 77 their urinary incontinence (UI) was not urge predominant, 19 had fewer than 7 episodes of incontinence per week and the other 38 were excluded for a variety of reasons.
Groups:
- Combination Therapy: Women randomly assigned to this condition receive 10 weeks of anti-cholinergic medication and behavioral training.
- Drug Therapy Alone: Women assigned to this arm received 10 weeks of anti-cholinergic medication, only.
Period: Baseline to 10 Weeks
Arm/Group | Combination Therapy | Drug Therapy Alone
Started | 154 | 153
Completed | 139 | 141
Not Completed | 15 | 12
Not completed — Lost to Follow-up | 15 | 12
Period: Baseline to 8 Months
Arm/Group | Combination Therapy | Drug Therapy Alone
Started | 154 | 153
Completed | 110 | 112
Not Completed | 44 | 41
Not completed — Lost to Follow-up | 44 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy | Drug Therapy Alone | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 106 | 218
  >=65 years | 42 | 47 | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (14.2) | 58.0 (13.5) | 56.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 153 | 307
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 154 | 153 | 307

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women Who Meet Definition of Success
Description: Proportion of women who meet definition of success: not taking drug or receiving other urge UI therapy (i.e., neuromodulation, botox injections, myomectomy, electrical stimulation, or any intravesical therapy) and not taking a tricyclic antidepressant or duloxetine at 8 months; and a >70% reduction in number of incontinence episodes as compared to baseline.
Time Frame: 8 months
Population: All women who completed the 8 months assessment or were known to return to drug use prior to that time.
Measure: Number; unit: participants
Arm/Group | Combination Therapy | Drug Therapy Alone
Number analyzed (Participants) | 118 | 119
participants | 43 | 41
Statistical Analysis 1: Comparison: Combination Therapy vs Drug Therapy Alone; Kaplan Meier Lifetable analysis was used to compute the 8 month cumulative success rates; Test type: Superiority or Other; p = 0.74, Log Rank; Difference in cumulative success rates = 0, 95% CI 2-sided [-0.12 to 0.12], Standard Error of Mean 0.06

2. Secondary Outcome: Change in Incontinence Episodes
Description: Change from baseline to 10 weeks in number of incontinence episodes per week as reported on bladder diary.
Time Frame: Baseline and 10 weeks
Population: All women with valid bladder diary at baseline and 10 weeks in each treatment group.
Measure: Mean (Standard Error); unit: incontinence episodes per week
Arm/Group | Combination Therapy | Drug Therapy Alone
Number analyzed (Participants) | 133 | 136
incontinence episodes per week | -20.4 (1.4) | -18.5 (1.4)
Statistical Analysis 1: Comparison: Combination Therapy vs Drug Therapy Alone; Test of hypothesis of no difference in change in episodes between the two groups; Test type: Superiority or Other; p = 0.34, ANOVA — Mixed effect repeated measures analysis of variance controlling for study site; Mean Difference (Net) = 1.9, 95% CI 2-sided [-2.0 to 5.9], Standard Error of Mean 2.0

3. Secondary Outcome: Change in Voids Per Day
Description: Change from baseline to 10 weeks in frequency of voids per day as reported on bladder diary
Time Frame: baseline and 10 weeks
Population: All women with valid bladder diary at baseline and 10 weeks in each treatment group.
Measure: Mean (Standard Error); unit: voids per day
Arm/Group | Combination Therapy | Drug Therapy Alone
Number analyzed (Participants) | 133 | 136
voids per day | -0.5 (0.4) | 0.3 (0.3)
Statistical Analysis 1: Comparison: Combination Therapy vs Drug Therapy Alone; Null hypothesis of no difference between arms in change in number of voids per day from baseline to 10 weeks; Test type: Superiority or Other; p = 0.08, ANOVA — Repeated measures ANOVA controlling for clinical site; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.7 to 0.1], Standard Error of Mean 0.5 — Difference (group 1 - group 2) in change from baseline to follow-up in voids per day

4. Secondary Outcome: Symptom Distress
Description: Urogenital distress inventory (UDI). Higher score indicates greater distress. Possible range 0 to 300.
Time Frame: baseline, 10 weeks and 8 months
Population: All women who completed UDI at each time in each treatment group
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combination at Baseline: Baseline value for women in combination therapy
- Combination at 10 Weeks: 10 week value for women in combination arm
- Combiniation at 8 Months: 8 months value from women in combination arm
- Drug Only at Baseline: Baseline value for women randomized to drug only
- Drug Only at 10 Weeks: 10 week value for women randomized to drug only
- Drug Only at 8 Months: 8 month value for women randomized to drug only
Arm/Group | Combination at Baseline | Combination at 10 Weeks | Combiniation at 8 Months | Drug Only at Baseline | Drug Only at 10 Weeks | Drug Only at 8 Months
Number analyzed (Participants) | 154 | 133 | 109 | 153 | 136 | 111
units on a scale | 121.4 (3.8) | 47.3 (4.1) | 61.9 (4.3) | 118.2 (3.9) | 58.1 (4.0) | 83.3 (4.2)
Statistical Analysis 1: Comparison: Combination at Baseline vs Combination at 10 Weeks vs Combiniation at 8 Months vs Drug Only at Baseline vs Drug Only at 10 Weeks vs Drug Only at 8 Months; Null hypothesis is that there is no difference between treatment groups in improvement in UDI over time; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — Repeated measures ANOVA; Main hypothesis tested by F-test for treatment by time interaction (2 and 509 degrees of freedom). No parameters estimated; Other = 0

5. Secondary Outcome: Symptom Bother
Description: Disease specific overactive bladder scale (OAB-q). HIgher score indicates greater bother. Possible range 0 to 100.
Time Frame: baseline, 10 weeks and 8 months
Population: Participants who completed OAB-q assessment at each time in each treatment group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination at Baseline | Combination at 10 Weeks | Combiniation at 8 Months | Drug Only at Baseline | Drug Only at 10 Weeks | Drug Only at 8 Months
Number analyzed (Participants) | 154 | 133 | 109 | 153 | 136 | 111
units on a scale | 59.9 (1.7) | 23.1 (1.8) | 29.0 (1.9) | 60.0 (1.7) | 29.6 (1.7) | 39.6 (1.8)
Statistical Analysis 1: Comparison: Combination at Baseline vs Combination at 10 Weeks vs Combiniation at 8 Months vs Drug Only at Baseline vs Drug Only at 10 Weeks vs Drug Only at 8 Months; Repeated measures analysis of difference in symptom bother over time by treatment group; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis — P-value for test of time by treatment group interaction; Adjusted for study site; Other = 0

6. Secondary Outcome: Satisfaction
Description: Number of women who responded "completely satisfied" to question, "How satisfied are you with your progress?"
Time Frame: 10 weeks
Population: Number of women who completed satisfaction question at 10 weeks.
Measure: Number; unit: participants
Arm/Group | Combination at 10 Weeks | Drug Only at 10 Weeks
Number analyzed (Participants) | 134 | 138
participants | 71 | 55
Statistical Analysis 1: Comparison: Combination at 10 Weeks vs Drug Only at 10 Weeks; Null hypothesis: no difference in satisfaction at 10 weeks; Test type: Superiority or Other; p = 0.02, Regression, Logistic; Controlling for clinical site and randomization stratum; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.09 to 2.92] — Ratio of odds of complete satisfaction in Combination therapy arm to Drug only arm

7. Secondary Outcome: Satisfaction
Description: Number of women who responded "completely satisfied" to question "How satisfied are you with your progress?"
Time Frame: 8 months
Population: Number of participants who completed the 8 months satisfaction questions
Measure: Number; unit: participants
Arm/Group | Combination Therapy | Drug Therapy Alone
Number analyzed (Participants) | 115 | 123
participants | 38 | 25
Statistical Analysis 1: Comparison: Combination Therapy vs Drug Therapy Alone; Null hypothesis: No difference in satisfaction at 8 months post intervention; Test type: Superiority or Other; p = 0.02, Regression, Logistic; Controlling for clinical site and randomization stratum; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.11 to 3.70] — Ratio of odds of complete satisfaction in combination therapy group compared to drug only group

8. Secondary Outcome: Symptom Improvement
Description: Number of women who responded "much better" or "better" to question: "Overall, do you feel that you are much better, better, about the same, worse or much worse?"
Time Frame: 10 weeks
Population: Participants who completed the satisfaction item at 10 weeks.
Measure: Number; unit: participants
Arm/Group | Combination Therapy | Drug Therapy Alone
Number analyzed (Participants) | 134 | 138
participants | 120 | 106
Statistical Analysis 1: Comparison: Combination Therapy vs Drug Therapy Alone; Null hypothesis: No difference in perceived improvement between women in combination therapy group compared to those in drug only group; Test type: Superiority or Other; p = 0.008, Regression, Logistic — P-value from logistic regression analysis; Controlling for clinical site and randomization stratum; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.27 to 5.13]

9. Secondary Outcome: Symptom Improvement
Description: as for outcome 8
Time Frame: 8 months
Population: Participants who completed the perceived improvement item at 8 months.
Measure: Number; unit: participants
Arm/Group | Combination Therapy | Drug Therapy Alone
Number analyzed (Participants) | 116 | 125
participants | 80 | 54
Statistical Analysis 1: Comparison: Combination Therapy vs Drug Therapy Alone; Null hypothesis: No difference in perceived improvement at 8 months between women in combination therapy group compared to those in drug only group; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Controlling for clinical site and randomization stratum; Odds Ratio (OR) = 3.17, 95% CI 2-sided [1.83 to 5.52]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events throughout the study period (8 months).
Arm/Group | Combination Therapy | Drug Therapy Alone
Serious Adverse Events (participants affected / at risk) | 2/154 | 2/153
Other Adverse Events (participants affected / at risk) | 2/154 | 1/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=154) | Drug Therapy Alone (N=153)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Small bowl obstruction (Gastrointestinal disorders) | 1 (2) | 1 (1)
Renal cell carcinoma (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=154) | Drug Therapy Alone (N=153)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Peripheral edema (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncopal episode (Cardiac disorders) | 1 (1) | 0 (0)
Night sweats (Renal and urinary disorders) | 1 (1) | 0 (0)
Stomach cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Ony 68% of participants completed assigned treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No